CLINICAL TRIAL: NCT04799509
Title: Assessment of the 90-day Mortality Risk Score After Video-assisted Thoracoscopic Lobectomy in the Italian VATS Group Cohort
Brief Title: Assessment of the 90-day Mortality Risk Score After VATS Lobectomy
Status: Completed | Type: Observational
Sponsor: Università degli Studi dell'Insubria (Other)
Responsible Party: Principal Investigator, Maria Cattoni, Principal Investigator - Clinician at Center for Thoracic Surgery - School of Medicine and Surgery - University of Insubria - Varese, Università degli Studi dell'Insubria
Other Study IDs: VALIDATION
Record Dates: First submitted 2021-03-12; First posted 2021-03-16 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Lung Cancer; Surgery--Complications; Morality
Keywords: non-small cell lung cancer; VATS lobectomy; 90-day postoperative mortality; risk score; validation
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: VATS lobectomy — VATS lobectomy

SUMMARY:
A five classes (A-E) aggregate risk score predicting 90-day mortality after video-assisted thoracoscopic lobectomy for lung cancer, including as independent factors male sex (3 points), carbon monoxide lung diffusion capacity <60% (1 point) and operative time >150 minutes (1 point), has been recently published. This study aims to assess the effectiveness and reliability of this risk model in a large, independent cohort of patients, in order to confirm its generalizability.

DETAILED DESCRIPTION:
From the Italian VATS Group Database, we selected patients who underwent video-assisted thoracoscopic lobectomy for non-small cell lung cancer. We calculated the aggregate risk score and the corresponding class of 90-day mortality risk for each patient. The correlation between risk classes and mortality rates was tested by Spearman's rho-test. Model calibration was evaluated by Hosmer-Lemeshow goodness-of-fit test.

ELIGIBILITY:
Inclusion Criteria:

- Patients undergoing VATS lobectomy for non-small cell lung cancer

Exclusion Criteria:

* Incomplete data for risk score calculation
* Tumor size >5 cm
* Follow-up <3 months
* Patients undergoing neoadjuvant treatment
* Patients undergoing extended resection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients were selected from the Italian VATS Group registry (a database containing prospectively collected data on VATS anatomical lung resection performed in 58 certified thoracic surgery centers from January 1st 2014). The VATS Group database was awarded by the European Society of Thoracic Surgeons in the 2017
Sampling Method: Probability Sample
Enrollment: 2209 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2018-11-27 (Actual); Study Completion 2018-11-27 (Actual)

PRIMARY OUTCOMES:
90-day postoperative mortality | 90 day post surgical procedure
  Alive/Death (cause of death)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Imperatori, MD, Study Director — Università degli Studi dell'Insubria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brunelli A, Dinesh P, Woodcock-Shaw J, Littlechild D, Pompili C. Ninety-Day Mortality After Video-Assisted Thoracoscopic Lobectomy: Incidence and Risk Factors. Ann Thorac Surg. 2017 Sep;104(3):1020-1026. doi: 10.1016/j.athoracsur.2017.02.083. Epub 2017 Jun 1. PMID 28577845